CLINICAL TRIAL: NCT04530487
Title: A Pilot Study of Allogeneic Hematopoietic Stem Cell Transplantation for Pediatric and Adolescent-Young Adults Patients With High Risk Solid Tumors
Brief Title: Donor Stem Cell Transplant After Chemotherapy for the Treatment of Recurrent or Refractory High-Risk Solid Tumors in Pediatric and Adolescent-Young Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0496; NCI-2020-05879 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0496 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Desmoplastic Small Round Cell Tumor; Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Desmoplastic Small Round Cell Tumor; Recurrent Malignant Peripheral Nerve Sheath Tumor; Recurrent Malignant Solid Neoplasm; Recurrent Neuroblastoma; Recurrent Rhabdomyosarcoma; Refractory Desmoplastic Small Round Cell Tumor; Refractory Malignant Peripheral Nerve Sheath Tumor; Refractory Malignant Solid Neoplasm; Refractory Neuroblastoma; Refractory Rhabdomyosarcoma
MeSH Terms: conditions — Desmoplastic Small Round Cell Tumor; Neuroectodermal Tumors, Primitive, Peripheral; Neurofibrosarcoma; Neuroblastoma; Rhabdomyosarcoma | interventions — Stem Cell Transplantation; Cyclosporine; Cyclosporins; Etoposide; fludarabine phosphate; Antilymphocyte Serum; thymoglobulin; Melphalan; Mycophenolic Acid; Tacrolimus; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (conditioning regimen, HSCT) (Experimental): CONDITIONING REGIMEN: Patients receive thiotepa IV over 2-4 hours, etoposide IV over 60 minutes on days -8 to -6, melphalan IV over 20 minutes on days -5 and -4, and fludarabine phosphate IV over 1 hour on days -5 to -3 in the absence of disease progression or unacceptable toxicity. Patients receiving umbilical cord transplant also receive rabbit anti-thymocyte globulin IV on days -3 and -4.
  TRANSPLANT: Patients undergo HSCT on day 0.
  GVHD PROPHYLAXIS: Beginning day -2, patients receive tacrolimus or cyclosporine IV continuously until able to receive PO. Patients continue tacrolimus or cyclosporine PO to day 60 and tapered to day 100. Patients also receive mycophenolate mofetil PO or IV every 8 hours until day 40 and tapered to day 90.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclosporine; Drug: Etoposide; Drug: Fludarabine Phosphate; Biological: Lapine T-Lymphocyte Immune Globulin; Drug: Melphalan; Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Drug: Thiotepa

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HSCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Cyclosporine — Given IV and PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Cyclosporine Modified; Gengraf; Neoral; OL 27-400; Sandimmune; SangCya
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Biological: Lapine T-Lymphocyte Immune Globulin — Given IV
  Other Names: Anti-Thymocyte Globulin Rabbit; Grafalon; Rabbit Anti-Human Thymocyte Globulin (RATG); Rabbit Anti-Thymocyte Globulin; Rabbit Antithymocyte Globulin; Rabbit ATG; rATG; Thymoglobulin
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: CellCept; MMF
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Drug: Thiotepa — Given IV
  Other Names: 1,1'',1''''-Phosphinothioylidynetrisaziridine; Girostan; N,N'', N''''-Triethylenethiophosphoramide; Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312

SUMMARY:
This phase II trial investigates side effects and how well donor stem cell transplant after chemotherapy works in treating pediatric and adolescent-young adults with high-risk solid tumor that has come back (recurrent) or does not respond to treatment (refractory). Chemotherapy drugs, such as fludarabine, thiotepa, etoposide, melphalan, and rabbit anti-thymocyte globulin work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before a donor stem cell transplant helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. When the healthy stem cells from a donor are infused into a patient, they may help the patient's bone marrow make more healthy cells and platelets and may help destroy any remaining cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess tolerability of allogeneic hematopoietic stem cell transplantation (HCT) for patients with chemo-responsive recurrent/refractory solid tumors as defined by transplant-related mortality (TRM) at day 30 and the rate of grade III or higher organ toxicity (Bearman Regimen-Related Toxicities Scale) attributable to conditioning occurring within 30 days.

SECONDARY OBJECTIVES:

I. Assess median time to platelet and neutrophil engraftment. II. Assess incidence of acute graft-versus-host disease (aGVHD) by day 100. III. Assess incidence of chronic GVHD (cGVHD) at day 100 and one year. IV. Assess rate of grade II organ toxicity through day 100. V. Assess rate of graft failure (primary and secondary) through day 100. VI. Assess rate of infectious complications through day 100. VII. Assess progression free survival (PFS) at day 100,180 and 365. VIII. Assess cumulative incidence of relapse, overall survival (OS) at 100 days and 1 year.

OUTLINE:

CONDITIONING REGIMEN: Patients receive thiotepa intravenously (IV) over 2-4 hours and etoposide IV over 60 minutes on days -8 to -6, melphalan IV over 20 minutes on days -5 and -4, and fludarabine phosphate IV over 1 hour on days -5 to -3 in the absence of disease progression or unacceptable toxicity. Patients receiving umbilical cord transplant also receive rabbit anti-thymocyte globulin IV on days -4 and -3.

TRANSPLANT: Patients undergo HSCT on day 0.

GVHD PROPHYLAXIS: Beginning day -2, patients receive tacrolimus or cyclosporine IV continuously until able to receive orally (PO). Patients continue tacrolimus or cyclosporine PO to day 60 and tapered to day 100. Patients also receive mycophenolate mofetil PO or IV every 8 hours until day 40 and tapered to day 90.

After completion of HSCT, patients are followed up for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Pathological criteria, including malignant recurrent/refractory solid tumors. This would include:

  * Ewing's/peripheral primitive neuroectodermal tumor (PNET)
  * Malignant peripheral nerve sheath tumor, neurofibrosarcoma
  * Rhabdomyosarcoma
  * Neuroblastoma (patients who are ineligible for tandem autologous transplant or who are at least 3 months post autologous HCT)
  * Desmoplastic small round cell tumor (DSRCT)- both new diagnoses as well as recurrent/refractory disease
* Patients must have chemo-responsive disease, defined as; 30% or greater decrease in the tumor target lesions when compared to its pre-treatment evaluation. Patients with complete response will be eligible to participate
* Available suitable HCT donor
* Creatinine clearance or glomerular filtration rate (GFR) >= 50 ml/min/1.73m^2, and not requiring dialysis
* Diffusing capacity of lung for carbon monoxide (DLCO) (corrected for hemoglobin) >= 50% predicted. If unable to perform pulmonary function tests, then oxygen (O2) saturation >= 92% in room air
* Bilirubin =< 3 x upper limit of normal (ULN) and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 5 x for age (with the exception of isolated hyperbilirubinemia due to Gilbert's syndrome)
* DONOR: Matched related donor bone marrow (10 of 10 HLA alleles [HLA-A, B, C, DR, and DQ]. Matched related donor peripheral blood stem cell (PBSC) is allowed only if collection of bone marrow (BM) is not available or refused by parents/donor
* DONOR: Matched allogeneic umbilical cord blood (UCB): related

  * High-resolution matching at A,B, DRB1 (minimum 4/6)
  * KIR major histocompatibility complex (MHC) class 1 preferential mismatch (minimum 4/6)
* DONOR: Matched allogeneic umbilical cord blood: unrelated

  * High-resolution matching at A,B, DRB1 (minimum 4/6) •*KIR MHC class 1 preferential mismatch (minimum 4/6)

Exclusion Criteria:

* Lack of histocompatible suitable related donor/ graft source
* End-organ failure that precludes the ability to tolerate the transplant procedure, including conditioning regimen
* Renal failure requiring dialysis
* Congenital heart disease resulting in congestive heart failure
* Ventilatory failure: requires invasive mechanical ventilation
* Human immunodeficiency virus (HIV) infection
* Uncontrolled bacterial, viral, or fungal infections (currently taking medication yet clinical symptoms progress); stable, controlled disease with treatment is not an exclusion criteria
* A female of reproductive potential who is pregnant, planning to become pregnant during the study, or is nursing a child
* Any patient who does not fulfill the inclusion criteria listed above

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy S Connors, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to accrual from 8/19/2020 to 7/23/2024. Participants were referred for the study both internally and externally.
Groups:
- Allogeneic Stem Cell Transplant in High Risk Solid Tumors: Matched Allogeneic Umbilical Cord Donor - thiotepa, etoposide, mephalan, rabbit ATG conditioning; tacrolimus/cyclosporine and MMF - GVHD prophylaxis
Period: Overall Study
Arm/Group | Allogeneic Stem Cell Transplant in High Risk Solid Tumors
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic Stem Cell Transplant in High Risk Solid Tumors
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 12 [12 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Allogeneic HCT
Description: To assess tolerability of allogeneic HCT for patients with chemo-responsive recurrent/refractory solid tumors as defined by transplant-related mortality (TRM) at day 30
Time Frame: By day +30 after allogeneic HCT infusion
Population: No analysis was performed as insufficient patients were enrolled for statistically significant conclusions.
Arm/Group | Allogeneic Stem Cell Transplant in High Risk Solid Tumors
Number analyzed (Participants) | 0

2. Primary Outcome: Rate of Organ Toxicity
Description: The rate of grade III or higher organ toxicity (Bearman Regimen-Related Toxicities Scale)[1] attributable to conditioning occurring within 30 days.
Time Frame: By day +30 after allogeneic HCT infusion
Population: No analysis was performed as insufficient patients were enrolled for statistically significant conclusions.
Arm/Group | Allogeneic Stem Cell Transplant in High Risk Solid Tumors
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the start of preparative regimen up to D+100 the collection of adverse events will reflect the onset and resolution date and maximum grade
Arm/Group | Allogeneic Stem Cell Transplant in High Risk Solid Tumors
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Stem Cell Transplant in High Risk Solid Tumors (N=1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Creatinine Increase (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Generalized Edema (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestions-HHV6 (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Platelet count decrease (Investigations) | 1 (1)
Lung infection - Pneumonia (Infections and infestations) | 1 (1)
Respiratory, thoracic and mediastinal disorders-tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Tachycardia- intermittent (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT04530487/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT04530487/ICF_000.pdf